CLINICAL TRIAL: NCT01096706
Title: Effects of Urocortins on Forearm Arterial Blood Flow in Healthy Volunteers
Brief Title: Effects of Urocortins on Forearm Arterial Blood Flow in Healthy Volunteers (Protocol 3)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SV.Protocol 3
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Vascular Disease; Heart Disease
Keywords: Urocortin 2; Urocortin 3; Nitric Oxide; Plethysmography; Forearm blood flow; Vascular; Heart failure; endothelium; Cyclo-oxygenase pathway; EDHF
MeSH Terms: conditions — Vascular Diseases; Heart Diseases; Heart Failure | interventions — Substance P; Sodium Chloride; Fluconazole; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Nitric Oxide Clamp (Experimental): Forearm blood flow response to Urocortins 2, 3 and Substance P in the presence of Nitric Oxide clamp
  Interventions: Drug: NO clamp
- Saline Placebo (Placebo Comparator): Forearm blood flow response to Urocortin 2, Urocortin 3 and Substance P in the presence of saline placebo.
  Interventions: Drug: Saline
- Fluconazole (Experimental): Forearm blood flow response to Urocortin 2, Urocortin 3 and Substance P in the presence of intra-arterial Fluconazole.
  Interventions: Drug: Fluconazole
- Aspirin (Experimental): Forearm blood flow response to Urocortin 2, Urocortin 3 and Substance P in the presence of cyclooxygenase inhibition with Aspirin.
  Interventions: Drug: Aspirin
- Combined (Experimental): Forearm blood flow response to Urocortin 2, Urocortin 3 and Substance P in the presence of inhibition of cycloxygenase, EDHF and NO pathways with Aspirin, Fluconazole and NO clamp.
  Interventions: Drug: Combined

INTERVENTIONS:
Drug: NO clamp — After a 20 minute saline washout period, ascending doses of Urocortin 2, Urocortin 3 and substance P (doses as per Protocol 2) will be infused intra-arterially in the presence or the absence of the 'nitric oxide clamp' that will be commenced prior to the infusion of Urocortin 2, Urocortin 3 and substance P, and will be continued throughout the study.
  Baseline blood samples will be taken from both forearms at the start of the study for full blood count, cholesterol, glucose, renal function and t-PA and PAI-1 activity and antigen concentrations. Bilateral venous blood samples will be taken at baseline, immediately before the start of Ucn2/Ucn3 infusion and at the end of each dose of Ucn2/Ucn3 for subsequent calculation of net release of t-PA and PAI-1.
  Other Names: Forearm vascular study - Bilateral forearm blood flow will be measured at baseline and after each dose of Ucn 2, 3 and Substance P
  Arms: Nitric Oxide Clamp
Drug: Saline — After a 20 minute saline washout, incremental doses of Urocortin 2, Urocortin 3 and Substance P (in doses as per Protocol 2) will be infused in the presence of saline placebo.
  Baseline blood samples will be taken from both forearms at the start of the study for full blood count, cholesterol, glucose, renal function and t-PA and PAI-1 activity and antigen concentrations. Bilateral venous blood samples will be taken at baseline, immediately before the start of Ucn2/Ucn3 infusion and at the end of each dose of Ucn2/Ucn3 for subsequent calculation of net release of t-PA and PAI-1.
  Other Names: Forearm vascular study - Bilateral forearm blood flow will be measured at baseline and after each dose of Ucn 2, 3 and Substance P.
  Arms: Saline Placebo
Drug: Fluconazole — After a 20 minute saline washout period, ascending doses of Urocortin 2, Urocortin 3 and substance P (doses as per Protocol 2) will be infused intra-arterially in the presence of Fluconazole (which serves to inhibit the EDHF pathway) that will be commenced prior to the infusion of Urocortin 2, Urocortin 3 and substance P, and will be continued throughout the study.
  Baseline blood samples will be taken from both forearms at the start of the study for full blood count, cholesterol, glucose, renal function, plasma Ucn 2 and 3 and t-PA and PAI-1 activity and antigen concentrations. Bilateral venous blood samples will be taken at after the top dose of Ucn2/Ucn3 infusion and before and after each dose of Substance P for subsequent calculation of plasma Ucn 2/ Ucn 3 and net release of t-PA and PAI-1.
  Arms: Fluconazole
Drug: Aspirin — Oral Aspirin (600mg stat) will be administered 30 minutes before start of the study. After a 20 minute saline washout period, ascending doses of Urocortin 2, Urocortin 3 and substance P (doses as per Protocol 2) will be infused intra-arterially in the presence of saline.
  Baseline blood samples will be taken from both forearms at the start of the study for full blood count, cholesterol, glucose, renal function, plasma Ucn 2 and 3 and t-PA and PAI-1 activity and antigen concentrations. Bilateral venous blood samples will be taken at after the top dose of Ucn2/Ucn3 infusion and before and after each dose of Substance P for subsequent calculation of plasma Ucn 2/ Ucn 3 and net release of t-PA and PAI-1.
  Arms: Aspirin
Drug: Combined — Oral Aspirin (600mg stat) is administered 30 minutes before start of the study. After a 20 minute saline washout period, ascending doses of Urocortin 2, Urocortin 3 and substance P (doses as per Protocol 2) will be infused intra-arterially in the presence of the 'nitric oxide clamp' that will be commenced prior to the infusion of Urocortin 2, Urocortin 3 and substance P, and will be continued throughout the study. Intra-arterial Fluconazole is also commenced at the time of the Nitric oxide clamp.
  This serves to inhibit the cyclooxygenase, EDHF and NO pathways of endothelial vasodilatation.
  Blood samples are taken as per previous arms.
  Arms: Combined

SUMMARY:
Impairment of the heart's pumping capacity (heart failure) remains a major clinical problem with a poor prognosis and the search for novel treatments remains an important area of research.

Urocortins are proteins that appear to increase blood flow and heart pumping activity. There has been particular interest in the role of Urocortins 2 & 3 (subtypes of Urocortins) in heart failure.

In this study, we will examine the effects and mechanisms of Urocortins 2 & 3 on forearm blood flow and release of natural blood clot dissolving factors in the forearm circulation of healthy volunteers. In particular, we look at the endothelial mechanisms of vasodilatation of Urocortin 2 and 3.

In this study, we will look at the role of the lining of the blood vessel (endothelium) in response to urocortin types 2 and 3. We hypothesise that urocortins 2 & 3 act via the endothelium to cause dilatation of the blood vessels and release of tissue-plasminogen activating factor (blood clot dissolving factor). We also hypothesise that urocortins have a role in maintaining the normal baseline level of blood flow in forearm arteries. In addition to the above, we will also look at the effect of temporarily blocking the effect of urocortins, using a specially designed blocker drug (Astressin 2B).

Utilising the well-established technique of 'forearm venous occlusion plethysmography', we will be able to focus on the local effects of urocortins on arterial blood flow in forearm vessels, without affecting this system in the body as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 18 - 65 years (inclusive)

Exclusion Criteria:

* Lack of informed consent- Age <18 years > 65 years
* Current involvement in a clinical trial
* Severe or significant co-morbidity including bleeding diathesis, renal or hepatic failure
* Smoker
* History of anaemia
* Recent infective/inflammatory condition
* Recent blood donation (prior 3 months)
* Positive baseline urine test for drugs of abuse (including cannabinoids, benzodiazepines, opiates, cocaine and amphetamines)
* History of allergy to Aspirin

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow | 3 hours
  The difference between forearm blood flow in response to incremental doses of Ucn2, Ucn3 and Sub P in the presence vs absence of 'the nitric oxide clamp'

SECONDARY OUTCOMES:
Net t-PA release | 3 hours
  Net release of t-PA evoked by Ucn 2, Ucn 3 and Substance P, in the presence vs absence of a 'nitric oxide clamp'.

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, PhD FRCP, Principal Investigator — University of Edinburgh
Locations (1):
- Wellcome Trust Clinical Research Facility, Royal Infirmary of Edinburgh, Edinburgh, Mid Lothian, United Kingdom

REFERENCES:
- [Derived] Venkatasubramanian S, Griffiths ME, McLean SG, Miller MR, Luo R, Lang NN, Newby DE. Vascular effects of urocortins 2 and 3 in healthy volunteers. J Am Heart Assoc. 2013 Jan 31;2(1):e004267. doi: 10.1161/JAHA.112.004267. PMID 23525432